CLINICAL TRIAL: NCT01112202
Title: Effect of Dabigatran on Coagulation Parameters in Patients Undergoing Elective Orthopaedic Surgery
Brief Title: Effect of Dabigatran on Coagulation parameters-an ex Vivo Study
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Edelgard Lindhoff-Last, Department of Vascular Medicine, University Hospital Frankfurt
Other Study IDs: Dabi2010
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2010-04

CONDITIONS: Effect of Dabigatran in Laboratory Coagulation Parameters
Keywords: direct thrombin inhibitors; Dabigatran; Coagulation parameters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dabigatran represent a new class of promising anticoagulation agents. As an oral direct thrombin inhibitor it has been effective in preventing venous thromboembolism in patients undergoing elective orthopaedic surgery. This ex vivo study is undertaken to investigate the ex-vivo effects of Pradaxa® on different coagulation parameters.

DETAILED DESCRIPTION:
This mono-centric, open-label study is undertaken to validate the effects of Dabigatran on coagulation parameters in plasma samples of 70 patients after hip or knee replacement surgery treated with Dabigatran 150-220 mg/d. Plasma samples are obtained by blood collection before, after 2 hours and after 12-14 hours after Dabigatran dosing in steady state (on 3rd - 5th day).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y

Exclusion Criteria:

* Hemorrhagic disorder
* Liver disease
* Anemia
* Severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients after hip or knee replacement surgery treated with Dabigatran 150-220 mg/d
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt, Germany